CLINICAL TRIAL: NCT06443970
Title: Physiological Consequences of Low and High Flow Endotracheal Suctioning Devices in Intubated Preterm and Term Infants
Brief Title: Low and High Flow Suctioning in Intubated Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Rakesh Sahni, Professor of Pediatrics, Columbia University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAU9006
Record Dates: First submitted 2024-05-13; First posted 2024-06-05 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Failure
Keywords: cardiorespiratory disturbances; neonates; EXSALTA; Endotracheal Suctioning
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: In each group of study infants (open and closed ETT suctioning), the enrolled subjects will experience ETT suctioning with both methods, i.e. with ED and SCW suctioning systems. Each study infant will undergo two sequential suctioning procedures each day during the two-day study period. On day-1, the infant will be randomly assigned the ED or SCW suctioning device during the first maneuver and the devices will be alternated during the second maneuver. The suctioning device order will be reversed on study day-2 as shown in the study protocol below. In all each infant will have four suctioning maneuvers over two days, two each with ED and SCW suctioning devices.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Exsalta Device suctioning (Experimental)
  Interventions: Device: Exsalta Suction Device
- Coventional wall suctioning (Active Comparator)
  Interventions: Device: Exsalta Suction Device

INTERVENTIONS:
Device: Exsalta Suction Device — Low flow endotracheal suction device

SUMMARY:
Preterm and term intubuted infants in the NICU will undergo two sequential suctioning procedures: a new, FDA-approved suction device called EXSALTA (ED) and the standard conventional wall (SCW). The physiological consequences, i.e. changes in heart rate (HR), oxygen saturation (SpO2), cerebral oxygenation (C-rSO2), and cerebral fractional oxygen extraction (C-FOE) between ED and SCW ETT tracheal suctioning system in both open and closed catheter system settings will be evaluated using a randomized cross over design in preterm and term infants receiving mechanical ventilation via an ETT. This study will evaluate the hypothesis that there will be significantly lower variations in HR, SpO2, C-rSO2, and C-FOE during ETT suctioning with ED compared to SCW suctioning systems under both open and close ETT suction settings.

DETAILED DESCRIPTION:
Respiratory failure in neonates frequently requires mechanical ventilation through an endotracheal tube (ETT). The presence of an ETT inhibits the infant's intrinsic ability to clear endogenous lung secretions effectively with compromised glottic closure and impaired muccociliary function, and thus regular supportive suctioning of the ETT is essential. The benefits of patent airway are evident, but adverse effects may also result from suctioning which are especially deleterious in extremely preterm infants with immature pulmonary and systemic hemodynamic function. These adverse effects include transient hypoxemia and oxygen desaturation, vasovagal reactions, altered central and cerebral hemodynamics, atelectasis, pneumothorax, and mucosal damage. The cardiorespiratory instability during ETT suctioning is partially attributed to alveolar decruitment and loss of lung volume from disconnecting the ETT from the ventilator circuit and negative suction pressure. Maintenance of lung volume is essential to optimize gas exchange and prevent ventilator induced lung injury. The magnitude of lung volume loss is related to catheter size and applied suctioning pressure and flow, highlighting the complexity of interaction between suction technique, lung mechanics and disease state. In accordance with industry standard codes, a high flow rate is essential to ensure the rapid removal of fluid and secretions from the desired site and the standard conventional wall (SCW) suction outlets provide a minimum flow of approximately 85 liters per minute. Such high flows can lead to endotracheal suctioning-induced alveolar decruitment that may of significant clinical relevance. Recently, a low flow technology suction device EXSALTA (ED) for clearing ETT secretions in patients on ventilators has been approved by FDA. The device uses peristaltic action to move fluids from the patient to a collection canister at a fixed flow rate of 1.4 L/min and eliminates the uncontrolled flow of air from the patient's lungs. The user selects a desired pressure level that is independent of the flow rate, a feature unavailable with SCW wall suction equipment used at patient's bedside. This exceptional microprocessor-controlled tabletop suction device, available at any suction setting, reduces risk of negative pressures in the lungs to help prevent alveolar collapse and hypoxia associated with standard suctioning techniques. This study will examine the hypothesis that there will be significantly lower variations in heart rate (HR), oxygen saturation (SpO2), cerebral oxygenation (C-rSO2), and cerebral fractional oxygen extraction (c-FOE) with ED compared to SCW suction system during open or closed ETT suctioning. To test this hypothesis, the physiological consequences of two ETT suctioning systems in preterm and term infants will be evaluated using the following aims:

AIM 1. To compare the variations in HR (bpm), SpO2 (%), C-rSO2 (%), C-FOE (%) between ED and SCW suctioning systems during routine standard care open and closed ETT suctioning.

AIM II. To compare the incidence (episodes) of cardiorespiratory disturbances, i.e. bradycardia (HR<80 bpm) and/or hemoglobin oxygen desaturation (SpO2) < 80% for more than 10s during suctioning with ED and SCW suctioning system during routine standard care open and closed ETT suctioning.

ELIGIBILITY:
Inclusion Criteria:

* Preterm and term infants with birth weight more than 1000g receiving ETT suctioning

Exclusion Criteria:

* Infants with cyanotic congenital heart disease and cardiac rhythm disorders (arrythmias) will be excluded from the study.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in heart rate (HR) | Before suctioning (baseline) and up to 1-hour after suctioning
  Measured as beats per minute
Change in oxygen saturation (SpO2) | Before suctioning (baseline) and up to 1-hour after suctioning
  Measured as percent (%) change
Change in cerebral oxygenation (C-rSO2) | Before suctioning (baseline) and up to 1-hour after suctioning
  Measured as percent (%) change
Change in cerebral fractional oxygen extraction (c-FOE) | Before suctioning (baseline) and up to 1-hour after suctioning
  Measured as difference in SpO2 and C-rSO2 (%)

SECONDARY OUTCOMES:
Incidence of bradycardia | Before suctioning (baseline) and up to 1-hour after suctioning
  Count (episodes) of HR<80% for more than 10 sec
Incidence of hemoglobin oxygen desaturation | Before suctioning (baseline) and up to 1-hour after suctioning
  Count (episodes) of SpO2<80% for more than 10 sec

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Sahni, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No